CLINICAL TRIAL: NCT04990960
Title: Experimental Study About Efficacy Of Physiotherapy Treatment vs Self-treatment In Axillary Web Syndrome After Axillary Dissection In Breast Cancer
Brief Title: Experimental Study About Physiotherapy Treatment vs Self-treatment In Axillary Web Syndrome After Axillary Dissection
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ospedale "Carlo Poma" - Mantova (Other)
Responsible Party: Principal Investigator, Laura Mutti, Physiotherapist, Ospedale "Carlo Poma" - Mantova
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 78-2017-SPERIM_ALTRO-MN28
Record Dates: First submitted 2021-04-28; First posted 2021-08-05 (Actual); Last update posted 2021-08-05 (Actual); Status verified 2021-08

CONDITIONS: Breast Neoplasms
Keywords: Axillary Web Syndrome
MeSH Terms: conditions — Breast Neoplasms | interventions — Physical Therapy Modalities

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Physiotherapist (Active Comparator): The Physiotherapist worked on adhered breast scars, stiffness in neck and arm movements and actively worked on AWS cords with gentle extensions and / or energetic detachment maneuvers. No self-treatment methods were offered and required of the subject.
  Interventions: Other: Physiotherapy
- Self-treatment (Experimental): The Physiotherapist worked on adhered breast scars, stiffness in neck and arm movements. During each session the patient was also assessed and trained in self-treatment exercises assigned to treat their cords. Subjects were trained to perform self-treatment extension exercises with four exercises selected by the Physiotherapist
  Interventions: Other: Physiotherapy

INTERVENTIONS:
Other: Physiotherapy — During each session (45 minutes)the patient was assessed and trained in self-treatment exercises assigned to treat their cords. This later method was chosen to ensure regular participation in their exercises and early correction of any inaccuracies in the implementation of the exercises regarding AWS treatment . Or the Physiotherapist worked actively on cords with soft or vigorous stretching.
  Other Names: Selftreatment

SUMMARY:
BACKGROUND Dissection and removal of Lymph nodes in the Axilla (ALND) remains a method used in breast cancer management across the world. Post- surgical scar tissue that forms in this dissection is therefore beyond the linear scar, is characterized by less elasticity than healthy tissue and can over time, because of the anatomical location, cause significant limitations of the Active Range of Motion (AROM) of the scapulohumeral joint. After this procedure it's possible that Axillary Web Syndrome (AWS) occurs. This study discusses the physiotherapy management of patients with AWS. The primary objective of the study was to verify direct and indirect changes to AWS cords with two treatment methods at a single breast cancer rehabilitation setting: Physiotherapist 's work Vs. Self-treatment.

DETAILED DESCRIPTION:
Breast cancer is the most common form of cancer among women. Axillary surgical procedures have reported, with post-operative morbidity of bleeding, lymphedema and shoulder pain, also the rather underestimated Axillary Web Syndrome. The study shows that the reduction of the problems linked to the Syndrome such as pain in shoulder Abduction and Flexion and inability in everyday life is possible with an early and competent treatment. Two different approaches to the Syndrome were investigated. The patients were divided in two groups. Good results were obtained within 5 weeks since the appearance of AWS with both of them but if the Physiotherapist is able to teach the convenient exercises, the selftreatment seemed to have the best outcome. This fact can change the awareness that an early approach is necessary inside the path to recovery. In the last years the Axillary Web Syndrome was the topic of many studies: the etiology, its clinical diagnosis, the relation with lymphedema…But the treatment was often reported like a combination of different techniques without indications about kinds, times. Instead the investigators examined a detailed procedure, the same in both groups. The work was different only as regards the cords treatment. This fact shows the value of a comprehensive treatment for neck, shoulder, breast and two different but specific works on the Axillary Web Syndrome. For these reasons its publishing could be important for all the professionals working with women after Surgery for breast cancer and metastatic lymphnodes.

ELIGIBILITY:
Inclusion Criteria:

1. Age > 18years;
2. Patients able to sign informed consent;
3. Patients who underwent ALND surgery for breast cancer;
4. Presence of cords associated with A.W.S.;
5. Surgeon examination carried no more than 10 days after the operation.

Exclusion Criteria:

1. Presence of cords after AD due to Melanoma metastasis.

Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 19 (Actual)
Dates: Start 2017-10-01 (Actual); Primary Completion 2019-09-30 (Actual); Study Completion 2019-10-30 (Actual)

PRIMARY OUTCOMES:
Average flexion | 5 weeks
  Starting position:the patient is laying on the table with the arm placed on the table and the hand opened touching the side with the palm (0° position).
  Flexion: the patient raises the arm towards the headboard (complete at 180°) The movements had been measured with a standard goniometer.

SECONDARY OUTCOMES:
Average abduction | 5 weeks
  Abduction: from the same start-position (0°), the patient moves the arm away from the leg (complete at 180°)

CONTACTS AND LOCATIONS:
Overall Officials: Laura Mutti, Principal Investigator — Hospital "Carlo Poma" - Mantova - Italy
Locations (1):
- Laura Mutti, Mantova, Italy

IPD SHARING:
Plan to Share IPD: No